CLINICAL TRIAL: NCT03771820
Title: Phase IIa/IIb Clinical Trial of NC-6004 in Combination With Pembrolizumab in Subjects With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck Who Have Failed Platinum or a Platinum-containing Regimen
Brief Title: Combination Therapy With NC-6004 and Pembrolizumab in Head and Neck Cancer Subjects Who Have Failed Platinum Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NanoCarrier Co., Ltd. (Industry)
Collaborators: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC-6004-009
Record Dates: First submitted 2018-11-01; First posted 2018-12-11 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: SCCHN
MeSH Terms: interventions — demplatin pegraglumer; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NC-6004 +pembrolizumab (Experimental): NC-6004 should be administered to subjects once every 3 weeks. On Day 1 of each treatment cycle NC-6004 will be administered first followed by pembrolizumab.
  In phase IIa portion, NC-6004 dose goes up from 90 mg/m2 up to 135 mg/m2. In phase IIb portion, the dose should be the determined RPII dose in phase IIa portion.
  Interventions: Drug: NC-6004; Drug: Pembrolizumab
- Pembrolizumab (Active Comparator): The recommended dose of pembrolizumab is 200 mg administered as an IV infusion over 30 minutes every 3 weeks.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: NC-6004 — NC-6004 should be administered to subjects once every 3 weeks. On Day 1 of each treatment cycle NC-6004 will be administered first followed by pembrolizumab.
  Other Names: Nanoplatin
  Arms: NC-6004 +pembrolizumab
Drug: Pembrolizumab — The recommended dose of pembrolizumab is 200 mg administered as an IV infusion over 30 minutes every 3 weeks.
  Other Names: Keytruda

SUMMARY:
In Phase IIa, dose-escalation study to determine the optimum tolerated dose and a recommended Phase IIb (RPIIb) dose in combination with pembrolizumab in subjects with recurrent or metastatic squamous cell carcinoma of the head and neck who have failed platinum or a platinum containing regimen.

In Phase IIb, randomized control study between NC-6004 in combination with pembrolizumab versus pembrolizumab alone in the same subject population as Part 1 at the RPIIb dose identified in PIIa.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Males or females aged ≥18 years at screening.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Have histologically- or cytologically-confirmed HNSCC.
* Have recurrent disease not amenable to curative treatment with local or systemic therapy, or metastatic (disseminated) HNSCC of the oral cavity, oropharynx, hypopharynx, or larynx that is considered incurable by local therapies.
* Having prior platinum failure.

Exclusion Criteria:

* Subjects with carcinoma of the nasopharynx, squamous cell carcinoma of unknown primary origination, squamous cell carcinoma that originates from the skin and salivary gland or paranasal sinus, nonsquamous histologies.
* Have disease that is suitable for locoregional treatment administered with curative intent or refuses curative intent.
* Have no more than 15% body weight loss due to the underlying condition in the last 3 months from signing of informed consent in Part 1 of the study and from randomization in to Part 2.
* Are currently participating in or have participated in a study of an investigational agent or are using an investigational device within 4 weeks prior to the first dose of trial treatment.
* Were previously treated with 3 or more lines of systemic therapies administered for recurrent and/or metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Determine the Recommended Phase (RPII) dose (mg/m2) of NC-6004 in combination with pembrolizumab | 1 year
  In PIIa portion, to determine RPII dose of NC-6004 in combination with pembrolizumab
Compare median Progression Free Survival (PFS) between NC-6004 +pembrolizumab and pembrolizumab alone | 1 year
  In PIIb portion, to compare PFS between NC-6004 plus pembrolizumab and pembrolizumab alone.

SECONDARY OUTCOMES:
Compare median Overall Survival (OS) between NC-6004 +pembrolizumab and pembrolizumab alone | 2 years
  In PIIb portion, to compare OS rate between NC-6004 plus pembrolizumab and pembrolizumab alone.
Compare overall response (complete response and partial response) rate between NC-6004 +pembrolizumab and pembrolizumab alone | 1 year
  In PIIb portion, to ORR between NC-6004 plus pembrolizumab and pembrolizumab alone
Compare duration of response between NC-6004 +pembrolizumab and pembrolizumab alone | 1 year
  In PIIb portion, to compare DOR between NC-6004 plus pembrolizumab and pembrolizumab alone
Compare time to response between NC-6004 +pembrolizumab and pembrolizumab alone | 1 year
  In PIIb portion, to compare TTR between NC-6004 plus pembrolizumab and pembrolizumab alone
Safety and tolerability as measured by severity of Adverse Events (AEs) | 1 year
  The safety endpoints for this study are the incidence and severity of AEs in accordance with the NCI CTCAE and the occurrence of SAEs and treatment discontinuations due to AEs
Assess the Maximum Plasma Concentration (Cmax) of NC-6004 in combination with pembrolizumab | 1 year
  Assess PK parameters of the Maximum Plasma Concentration (Cmax)
Assess the Time to Maximum Concentration (Tmax) of NC-6004 in combination with pembrolizumab | 1 year
  Assess PK parameters of Time to Maximum Concentration (Tmax)
Assess the Area Under the Concentration (AUC) of NC-6004 in combination with pembrolizumab | 1 year
  Assess PK parameters of Area Under the Concentration (AUC)
Assess the Half-life(T½) of NC-6004 in combination with pembrolizumab | 1 year
  Assess PK parameters of Half-life(T½)
Assess the Clearance (CL) of NC-6004 in combination with pembrolizumab | 1 year
  Assess PK parameters of Clearance (CL)
Assess the Volume of Distribution (V) of NC-6004 in combination with pembrolizumab | 1 year
  Assess PK parameters of Volume of Distribution (V)

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Osada, Study Director — NanoCarrier US LLC
Locations (24):
- Croatia (3):
  - 0603, Osijek
  - 0601, Zagreb
  - 0602, Zagreb
- Czechia (3):
  - 0701, Brno
  - 0702, Hradec Králové
  - 0703, Olomouc
- Hungary (4):
  - 0104, Budapest
  - 0105, Debrecen
  - 0103, Kecskemét
  - 0101, Pécs
- Poland (2):
  - 0202, Bydgoszcz
  - 0201, Lodz
- Russia (2):
  - 0802, Omsk
  - 0801, Yekaterinburg
- Serbia (3):
  - 0301, Belgrade
  - 0301, Kamenitz
  - 0303, Niš
- Taiwan (4):
  - 0404, Taichung
  - 0402, Taipei
  - 0403, Taipei
  - 0401, Taoyuan
- Ukraine (3):
  - 0902, Cherkasy
  - 0903, Ivano-Frankivsk
  - 0904, Kharkiv

IPD SHARING:
Plan to Share IPD: Undecided